CLINICAL TRIAL: NCT03718416
Title: Non-Interventional, Observational, Natural History Study of Serious Medical Events in Prader-Willi Syndrome
Brief Title: Natural History Study of Serious Medical Events in PWS
Acronym: PATH for PWS
Status: Completed | Type: Observational
Sponsor: Foundation for Prader-Willi Research (Other)
Collaborators: Prader-Willi Syndrome Association USA (Other); Foundation for Prader-Willi Research Canada (Unknown); Prader-Willi Research Foundation Australia (Unknown); Prader-Willi Syndrome Association (Other)
Responsible Party: Sponsor
Other Study IDs: PATH-PWS-001
Record Dates: First submitted 2018-10-12; First posted 2018-10-24 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Prader-Willi Syndrome
Keywords: observational; non-interventional; Prader-Willi syndrome; PWS
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PATH for PWS is a study to help researchers better understand serious medical events in PWS over a 4-year period, as well as evaluate how PWS-related behaviors change over time. The data from this study is intended to inform the development and clinical trial design of potential new treatments.

DETAILED DESCRIPTION:
Every 6 months, participants or their caregivers will be asked to update online surveys about medical problems and serious medical events, as well as provide information about conditions and behaviors often associated with PWS such as hyperphagia. Because this is an observational study, no study drug will be provided and no visits to a doctor or clinic are required.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

* Confirmed diagnosis of PWS
* At least 5 years of age
* Live in the United States, Canada, Australia, or New Zealand
* Must be enrolled or willing to enroll in the Global PWS Registry (https://pwsregistry.org)

Participants or their caregiver must also meet all of the following criteria:

* Have access to the internet to complete online surveys at least every 6 months
* Agree to receive reminders to complete online surveys
* Allow the staff to ask questions about survey responses if more information is needed and to enter data into the surveys

Exclusion Criteria:

Participants or their caregiver meeting any of the following criteria will be excluded:

* Is not able to read and understand English

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with PWS who are at least 5 years old and live in the United States, Canada, Australia, or New Zealand
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the incidence of serious medical events | Up to 4 years
  Serious medical events are those that result in death, are life-threatening, require hospitalization or an emergency room visit, or are medically significant

SECONDARY OUTCOMES:
Evaluate the incidence of non-serious thrombotic events | Up to 4 years
  Thrombotic events include blood clots in a blood vessel, such as an artery or vein
Analyze D-dimer concentrations in a subset of participants who agree to provide a blood sample | Up to 4 years
  D-dimer is a protein in the blood that is present when a blood clot is forming or has formed
Evaluate prescription medication use associated with serious medical events and thrombotic events | Up to 4 years
Evaluate the change in weight | Up to 4 years
Evaluate the change in height | Up to 4 years
Evaluate the change in height-adjusted weight | Up to 4 years
Evaluate PWS complexity using an online survey | Up to 4 years
Evaluate the pattern of hyperphagia behaviors using an online survey | Up to 4 years
  Hyperphagia means the intense, constant hunger that often occurs in individuals with PWS
Evaluate hyperphagia management using an online survey | Up to 4 years
Evaluate food-related behaviors using an online survey | Up to 4 years
Analyze medical information to evaluate the natural history of PWS | Up to 4 years
  Medical information will be from birth to before enrolling in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation for Prader-Willi Research (FPWR), Walnut, California, United States

IPD SHARING:
Plan to Share IPD: Yes
FPWR allows for registry use by request and releases de-identified data to the public.
Access Criteria: Data access will be governed by the Global PWS Registry advisory board.

REFERENCES:
- [Derived] Strong TV, Miller JL, McCandless SE, Gevers E, Yanovski JA, Matesevac L, Bohonowych J, Ballal S, Yen K, Hirano P, Cowen NM, Bhatnagar A. Behavioral changes in patients with Prader-Willi syndrome receiving diazoxide choline extended-release tablets compared to the PATH for PWS natural history study. J Neurodev Disord. 2024 Apr 26;16(1):22. doi: 10.1186/s11689-024-09536-x. PMID 38671361
- See also: Global Prader-Willi Syndrome Registry — https://pwsregistry.org/
- See also: Foundation for Prader-Willi Research Website — https://www.fpwr.org/
- See also: PATH for PWS / PATH-PWS-001 Study Website — https://www.pathforpws.com